CLINICAL TRIAL: NCT00306735
Title: A Double-blind Phase 2 Study to Assess the Safety and Efficacy of Aloxi (Palonosetron HCl) for the Prevention of Nausea and Vomiting in Multiple Myeloma Patients Receiving High-dose Melphalan as Conditioning Chemotherapy for Stem Cell Transplantation
Brief Title: Safety and Efficacy Study for the Prevention of Nausea and Vomiting in Multiple Myeloma Patients Receiving Stem Cell Transplantation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Helsinn Healthcare SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PALO-05-05
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Stem Cell Transplantation; CINV
MeSH Terms: conditions — Multiple Myeloma | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palonosetron (Experimental)
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron

SUMMARY:
The primary purpose of this study is to explore the efficacy of three different dose schedules of palonosetron for the prevention of emesis over a 7-day study interval in multiple myeloma patients.

DETAILED DESCRIPTION:
A number of multiple-day chemotherapy regimens involving moderately or highly emetogenic agents are used for the treatment of cancers. Further, patients undergoing high-dose conditioning regimens in combination with bone marrow or stem cell transplants remain poorly controlled in terms of CINV. Patients treated with these regimens are at risk for developing CINV with each treatment as well as in the delayed setting.

Palonosetron to date, has been studied against single-day moderately and highly emetogenic chemotherapy regimens. It is of interest, therefore, to explore the safety and efficacy of palonosetron when administered during a multiple-day chemotherapy regimen. For this purpose, a population receiving melphalan (100 mg/m^2) as a conditioning regimen before stem cell transplant for the treatment of multiple myeloma was selected.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age greater than or equal to 18 years
3. Histologically confirmed multiple myeloma
4. Karnofsky index greater than or equal to 50%
5. Scheduled to receive a regimen containing melphalan at a dose of 100 mg/m^2 on Study Days -2 and -1 followed by autologous stem cell transplant on Day 0
6. Known mild to moderate hepatic, renal or cardiovascular impairment may be enrolled at the discretion of the investigator
7. Women of childbearing potential must use reliable contraceptive measures and have negative pregnancy tests at screening

Exclusion Criteria:

1. Inability or unwillingness to understand or to cooperate with the study procedures
2. Received any investigational drugs within 30 days before study entry
3. Received any drug with potential antiemetic efficacy within 24 hours prior to the start of chemotherapy on Study Day -2 or are scheduled to receive or anticipate use of any drug of this type (with the exception of palonosetron or dexamethasone as indicated for this study) during the trial, including the following:

   1. 5-HT3 receptor antagonists;
   2. Dopamine receptor antagonists (metoclopramide);
   3. Phenothiazine antiemetics (prochlorperazine, thiethylperazine and perphenazine);
   4. Atypical antipsychotic agents with Compazine-like activity (e.g. olanzapine, risperidone);
   5. Haloperidol, droperidol, tetrahydrocannabinol, or nabilone;
   6. Any systemic corticosteroid (hydrocortisone, methylprednisolone, prednisone), unless used as a preventative measure for chemotherapy toxicities. Topical or inhaled preparations are allowed; and,
   7. Any non-prescription medication, nutritional supplements, vitamins or herbal-type products known to either cause nausea or vomiting or used to treat nausea or vomiting.

   Note: with the exception of first-generation 5-HT3-receptor antagonists, above medication(s) may be used as rescue medication.
4. Any vomiting, retching or National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version 3.0, Grade 2-4 nausea in the 24 hours preceding chemotherapy;
5. Ongoing vomiting for any organic etiology;
6. Scheduled to receive any other emetogenic chemotherapeutic agents during the study other than those specified in the protocol;
7. Known contraindication to 5-HT3 receptor antagonists;
8. Received, or will receive, radiotherapy of upper abdomen or cranium or total body irradiation within one week prior to or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schuster, M.D., Principal Investigator — Cornell Medical Center, Division of Hematology-Oncology
Locations (10):
- United States (10):
  - Indiana Blood and Marrow Transplantation, Beech Grove, Indiana
  - Cornell Medical Center, New York, New York
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase-Temple, Philadelphia, Pennsylvania
  - Baylor University Blood and Marrow Transplantation, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fairfax-Northern Virginia Hematology-Oncology PC, Fairfax, Virginia